CLINICAL TRIAL: NCT01317615
Title: A Multi-centric, Open-label, Phase II Study Investigating the Combination of Afinitor With Paclitaxel and Carboplatin in First Line Treatment of Patients With Advanced (Stage IV) Large Cell Lung Cancer With Neuroendocrine Differentiation (LC-NEC)
Brief Title: RAD001 With Paclitaxel and Carboplatin in First Line Treatment of Patients With Advanced Large Cell Lung Cancer With Neuroendocrine Differentiation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRAD001KDE37; EudraCT 2010-022273-34 (Registry Identifier: EudraCT); 2010-022273-34
Record Dates: First submitted 2011-03-16; First posted 2011-03-17 (Estimated); Results first posted 2016-03-30 (Estimated); Last update posted 2016-03-30 (Estimated); Status verified 2016-02

CONDITIONS: Carcinoma, Large Cell; Neuroendocrine Tumors
Keywords: Large cell carcinoma,; Lung cancer,; Neuroendocrine Tumors,; RAD001
MeSH Terms: conditions — Carcinoma, Large Cell; Neuroendocrine Tumors; Lung Neoplasms | interventions — Everolimus; Paclitaxel; Carboplatin

ARMS (1):
- RAD001 plus paclitaxel/carboplatin (Experimental): Participants received RAD001 5 mg orally once daily in combination with carboplatin and paclitaxel for a maximum 4 cycles or until discontinuation.
  Interventions: Drug: RAD001; Drug: Paclitaxel; Drug: Carboplatin

INTERVENTIONS:
Drug: RAD001 — Participants started RAD001 treatment with a dose of 5 mg/day once daily. A dose decrease to 5 mg every other day was allowed if tolerability issues arose.
  Other Names: Everolimus
Drug: Paclitaxel — Paclitaxel was started at doses of 175 mg/m². Dose reductions of Paclitaxel to 135 mg/m2 was permitted if tolerability issues arose.
Drug: Carboplatin — Carboplatin was started at doses of Area under the Curve 5 (AUC 5). Dose reductions of carboplatin to AUC 4 was permitted if tolerability issues arose.

SUMMARY:
This is a multi-centric, open-label study evaluating the efficacy and safety of RAD001 in patients with advanced (stage IV) Lung Cancer (Large Cell) with neuroendocrine differentiation treated with a combination of RAD001 with paclitaxel and carboplatin.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who give a written informed consent obtained according to local guidelines
2. Histologically confirmed diagnosis of stage IV lung cancer of LC-NEC type according to WHO classification:

   1. Histolocial analysis of newly diagnosed disease must not be older than 8 weeks from signed consent
   2. Relapse must be confirmed by histology
   3. Neuroendocrine differentiation
3. World Health organisation (WHO) performance status grade ≤ 1
4. measurable disease
5. Adequate bone marrow function
6. Adequate liver function
7. Adequate renal function

Exclusion Criteria:

1. History or clinical evidence of central nervous system (CNS) metastases.
2. Presence of SCLC cells
3. Patients who have a history of another primary malignancy ≤ 3 years, with the exception of inactive basal or squamous cell carcinoma of the skin or cervical cancer in situ, early stages of breast cancer (LCIS and DCIS) and prostate cancer (stage T1a)
4. prior chemotherapy for the treatment of advanced lung cancer and/or not having recovered from the side effects of any other therapy (adjuvant treatment for earlier stages I-III is allowed if finished at least one year before study entry)
5. Patients who have received any investigational drug ≤ 28 days before starting study treatment or who have not recovered from side effects of such therapy
6. Patients who have not recovered from the side effects of any major surgery or patients that may require major surgery during the course of the study
7. Patients who have received prior therapy with RAD001 or other mTOR inhibitors
8. Having any severe and/or uncontrolled medical conditions
9. Women who are pregnant or breast feeding

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2011-04; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (9):
- Germany (9):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bremen
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Gauting
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Hemer
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Ulm

REFERENCES:
- [Derived] Christopoulos P, Engel-Riedel W, Grohe C, Kropf-Sanchen C, von Pawel J, Gutz S, Kollmeier J, Eberhardt W, Ukena D, Baum V, Nimmrich I, Sieder C, Schnabel PA, Serke M, Thomas M. Everolimus with paclitaxel and carboplatin as first-line treatment for metastatic large-cell neuroendocrine lung carcinoma: a multicenter phase II trial. Ann Oncol. 2017 Aug 1;28(8):1898-1902. doi: 10.1093/annonc/mdx268. PMID 28535181

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an open-label, single arm study.
Period: Overall Study
Arm/Group | RAD001 Plus Paclitaxel/Carboplatin
Started | 49
Completed | 0
Not Completed | 49
Not completed — Disease progression | 25
Not completed — New cancer therapy | 5
Not completed — Death | 6
Not completed — Withdrawal by Subject | 5
Not completed — Abnormal laboratory value(s) | 1
Not completed — Adverse Event | 7

BASELINE CHARACTERISTICS:
Arm/Group | RAD001 Plus Paclitaxel/Carboplatin
Number analyzed (Participants) | 49
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 35

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Progression-free
Description: Tumors were assessed according to Response Evaluation Criteria in Solid tumors (RECIST) to determine progression-free status. Complete response (CR): disappearance of all lesions (i.e. all evidence of disease, not just the target lesions) determined by 2 observations not less than 4 weeks apart; Partial response (PR): > 30% decrease in the sum of longest diameters of target lesions compared to baseline, with response or stable disease observed in non-target lesions, and no new lesions; Stable disease (SD): neither sufficient shrinkage to qualify for response or sufficient increase to qualify for progressive disease in target lesions, with response or stable disease observed in non-target lesions, and no new lesions; Progressive disease (PD): > 20% increase in the sum of longest diameters of target lesions compared to smallest sum longest diameter recorded. In addition, the sum must also demonstrate an absolute increase of at least 5mm.
Time Frame: 3 months
Population: All participants were included in the analysis.
Measure: Number; unit: Percentage of participants
Arm/Group | RAD001 Plus Paclitaxel/Carboplatin
Number analyzed (Participants) | 49
Percentage of participants | 49.0

2. Secondary Outcome: Percentage of Participants Progression-free
Description: Tumors were assessed according to Response Evaluation Criteria in Solid tumors (RECIST) to determine progression-free status. Complete response (CR) is disappearance of all lesions (i.e. all evidence of disease, not just the target lesions) determined by 2 observations not less than 4 weeks apart; Partial response (PR) is > 30% decrease in the sum of longest diameters of target lesions compared to baseline, with response or stable disease observed in non-target lesions, and no new lesions; Stable disease (SD) is neither sufficient shrinkage to qualify for response or sufficient increase to qualify for progressive disease in target lesions, with response or stable disease observed in non-target lesions, and no new lesions; and Progressive disease (PD is: > 20% increase in the sum of longest diameters of target lesions compared to smallest sum longest diameter recorded. In addition, the sum must also demonstrate an absolute increase of at least 5mm.
Time Frame: 6 months
Population: All participants were included in the analysis.
Measure: Number; unit: Percentage of participants
Arm/Group | RAD001 Plus Paclitaxel/Carboplatin
Number analyzed (Participants) | 49
Percentage of participants | 8.2

3. Secondary Outcome: Percentage of Participants With Overall Response Rate (ORR)
Description: ORR was defined as is the proportion of participants with a best overall response of CR or PR. CR is disappearance of all lesions (i.e. all evidence of disease, not just the target lesions) determined by 2 observations not less than 4 weeks apart; Partial response. PR is > 30% decrease in the sum of longest diameters of target lesions compared to baseline, with response or stable disease observed in non-target lesions, and no new lesions.
Time Frame: 3 months
Population: All participants were included in the analysis.
Measure: Number; unit: Percentage of participants
Arm/Group | RAD001 Plus Paclitaxel/Carboplatin
Number analyzed (Participants) | 49
Percentage of participants | 44.9

4. Secondary Outcome: Percentage of Participants With Disease Control Rate (DCR)
Description: DCR was defined as is the percentage of participants with a best overall response of CR or PR or SD. Complete response (CR) is disappearance of all lesions (i.e. all evidence of disease, not just the target lesions) determined by 2 observations not less than 4 weeks apart; Partial response (PR) is > 30% decrease in the sum of longest diameters of target lesions compared to baseline, with response or stable disease observed in non-target lesions, and no new lesions; Stable disease (SD) is neither sufficient shrinkage to qualify for response or sufficient increase to qualify for progressive disease in target lesions, with response or stable disease observed in non-target lesions, and no new lesions; and Progressive disease (PD is: > 20% increase in the sum of longest diameters of target lesions compared to smallest sum longest diameter recorded. In addition, the sum must also demonstrate an absolute increase of at least 5mm.
Time Frame: 3 months
Population: All participants were included in the analysis.
Measure: Number; unit: Percentage of participants
Arm/Group | RAD001 Plus Paclitaxel/Carboplatin
Number analyzed (Participants) | 49
Percentage of participants | 73.5

5. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as the time from the date of start of treatment to date of event defined as the first documented progression or death due to any cause.
Time Frame: 6 months
Population: All participants were included in the analysis.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | RAD001 Plus Paclitaxel/Carboplatin
Number analyzed (Participants) | 49
Days | 132 [97 to 181]

6. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from date of start of treatment to date of death due to any cause.
Time Frame: 12 months
Population: All participants were included in the analysis.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | RAD001 Plus Paclitaxel/Carboplatin
Number analyzed (Participants) | 49
Days | 298 [207 to 351]

ADVERSE EVENTS:
Arm/Group | RAD001 Plus Paclitaxel/Carboplatin
Serious Adverse Events (participants affected / at risk) | 28/49
Other Adverse Events (participants affected / at risk) | 43/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RAD001 Plus Paclitaxel/Carboplatin (N=49)
ANAEMIA (Blood and lymphatic system disorders) | 1
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 1
NEUTROPENIA (Blood and lymphatic system disorders) | 1
ATRIAL FIBRILLATION (Cardiac disorders) | 2
VERTIGO (Ear and labyrinth disorders) | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 1
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 2
COLITIS (Gastrointestinal disorders) | 1
CONSTIPATION (Gastrointestinal disorders) | 2
DIARRHOEA (Gastrointestinal disorders) | 1
GASTRITIS (Gastrointestinal disorders) | 1
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1
NAUSEA (Gastrointestinal disorders) | 1
FATIGUE (General disorders) | 1
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 5
MULTI-ORGAN FAILURE (General disorders) | 1
PAIN (General disorders) | 2
ACUTE HEPATIC FAILURE (Hepatobiliary disorders) | 1
HEPATOMEGALY (Hepatobiliary disorders) | 1
CLOSTRIDIAL INFECTION (Infections and infestations) | 1
EMPYEMA (Infections and infestations) | 1
EPIDIDYMITIS (Infections and infestations) | 1
GASTROENTERITIS (Infections and infestations) | 1
INFECTION (Infections and infestations) | 1
PNEUMONIA (Infections and infestations) | 3
PYOPNEUMOTHORAX (Infections and infestations) | 1
SEPSIS (Infections and infestations) | 2
SINUSITIS (Infections and infestations) | 1
C-REACTIVE PROTEIN INCREASED (Investigations) | 1
DEHYDRATION (Metabolism and nutrition disorders) | 2
HYPONATRAEMIA (Metabolism and nutrition disorders) | 2
PAIN IN JAW (Musculoskeletal and connective tissue disorders) | 1
SPINAL PAIN (Musculoskeletal and connective tissue disorders) | 1
BENIGN NEOPLASM OF THYROID GLAND (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
BRONCHIAL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
MALIGNANT NEOPLASM PROGRESSION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
METASTASES TO CENTRAL NERVOUS SYSTEM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
PARANEOPLASTIC SYNDROME (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
SCIATICA (Nervous system disorders) | 1
VOCAL CORD PARESIS (Nervous system disorders) | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 5
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 1
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 3
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 3
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | RAD001 Plus Paclitaxel/Carboplatin (N=49)
ANAEMIA (Blood and lymphatic system disorders) | 14
LEUKOPENIA (Blood and lymphatic system disorders) | 7
NEUTROPENIA (Blood and lymphatic system disorders) | 10
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 8
VISUAL IMPAIRMENT (Eye disorders) | 3
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 3
CONSTIPATION (Gastrointestinal disorders) | 9
DIARRHOEA (Gastrointestinal disorders) | 10
DYSPHAGIA (Gastrointestinal disorders) | 3
NAUSEA (Gastrointestinal disorders) | 13
STOMATITIS (Gastrointestinal disorders) | 8
ASTHENIA (General disorders) | 4
CHEST PAIN (General disorders) | 3
FATIGUE (General disorders) | 17
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 3
MUCOSAL INFLAMMATION (General disorders) | 8
OEDEMA PERIPHERAL (General disorders) | 7
PAIN (General disorders) | 6
PERIPHERAL SWELLING (General disorders) | 4
PYREXIA (General disorders) | 3
INFECTION (Infections and infestations) | 4
WEIGHT DECREASED (Investigations) | 8
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 3
DECREASED APPETITE (Metabolism and nutrition disorders) | 10
HYPOKALAEMIA (Metabolism and nutrition disorders) | 5
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 5
GROWING PAINS (Musculoskeletal and connective tissue disorders) | 3
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 3
HEADACHE (Nervous system disorders) | 6
HYPOAESTHESIA (Nervous system disorders) | 3
PARAESTHESIA (Nervous system disorders) | 7
POLYNEUROPATHY (Nervous system disorders) | 9
INSOMNIA (Psychiatric disorders) | 3
SLEEP DISORDER (Psychiatric disorders) | 5
COUGH (Respiratory, thoracic and mediastinal disorders) | 8
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 3
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 13
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 3
ALOPECIA (Skin and subcutaneous tissue disorders) | 12
NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 4
RASH (Skin and subcutaneous tissue disorders) | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.